CLINICAL TRIAL: NCT02982356
Title: Prenatal Screening, Diagnosis and Intrauterine Intervention of Fetal Abnormal Chromosome and Structure in Twins Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Collaborators: Children's Hospital of Fudan University (Other); International Peace Maternity and Child Health Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiFMIH-FMU2
Record Dates: First submitted 2016-11-29; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Chromosome Abnormality; Twin Pregnancy With Antenatal Problem
MeSH Terms: conditions — Chromosome Aberrations | interventions — Potassium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fetal Selective Reduction Technology (Other): Potassium chloride fetal heart injection in the dichorial twins with abnormal chromosome and structure
  Interventions: Procedure: Fetal Selective Reduction Technology; Drug: Potassium Chloride
- control group (No Intervention): normal dichorial twins without any intervention

INTERVENTIONS:
Procedure: Fetal Selective Reduction Technology — Fetal Selective Reduction Technology will be conducted according to different gestational weeks: before 16weeks, 16~24 weeks, 24~27+6 weeks,>28weeks
  Arms: Fetal Selective Reduction Technology
Drug: Potassium Chloride
  Arms: Fetal Selective Reduction Technology

SUMMARY:
The risk of abnormal chromosome and structure is much higher in twins than in singletons, and traditional early pregnancy screening strategy for single pregnancy is not suitable for twins. Based on our management experience of fetal medicine at twin pregnancy, and multi-center cooperation, the study will carry out the following clinical studies:

1. to explore a suitable, early, noninvasive and accurate prenatal screening strategy for twin pregnancy.
2. fetal chromosomal abnormalities

ELIGIBILITY:
Inclusion Criteria:

* ultrasound diagnosis as twin pregnancy
* at 11-14 gestational weeks

Exclusion Criteria:

* Multiple pregnancies (three or more)
* Maternal history of chromosome aneuploidy abnormality or tumor

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1300 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Success rate for the operation | 1 week

SECONDARY OUTCOMES:
long-term complications after surgery | 1 year

IPD SHARING:
Plan to Share IPD: Undecided
The Individual Participant Data sharing plan will be discussed with the other collaborators